CLINICAL TRIAL: NCT03937856
Title: Smartphone App Mindfulness-Based Intervention for Patients With Rheumatic Diseases
Brief Title: Smartphone Mindfulness Meditation for Patients With Rheumatic Diseases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving the institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00199546
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Inflammatory Arthritis; Scleroderma; Myositis; Sjogren's Syndrome; Systemic Lupus Erythematosus; Vasculitis
MeSH Terms: conditions — Arthritis; Scleroderma, Diffuse; Myositis; Sjogren's Syndrome; Lupus Erythematosus, Systemic; Vasculitis

STUDY DESIGN:
Intervention Model Description: Participants who choose the intervention arm will be asked to use the Calm application for 30 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participant groups will include enrolled patients with rheumatic disease who use the smartphone mindfulness meditation application for 30 days.
  Interventions: Behavioral: Calm- Mindfulness Meditation smartphone application
- Control group (No Intervention): Usual care participants.

INTERVENTIONS:
Behavioral: Calm- Mindfulness Meditation smartphone application — Participants will be asked to register and download the Calm application on participants' phones or home computer. Daily use for a minimum of 5 minutes will be suggested and will be recorded at study end.
  Arms: Intervention group

SUMMARY:
This study will assess the effect of a mindfulness meditation program administered via a smartphone application on health-related quality of life for patients with rheumatic disease.

DETAILED DESCRIPTION:
After obtaining written consent, participants will be asked to download and use the Calm meditation smartphone application everyday for a 30-day period. Participant demographics and clinical information will be collected at baseline. Participants will additionally be asked to complete questionnaires concerning health-related quality of life (HRQoL) as well as mental health, stress, and self-efficacy at baseline and at the end of the 30 day study period. A brief check-in via telephone will be conducted on day 15.

Participants using the calm app will be compared to participants receiving usual care who will be asked to complete identical sets of questionnaires. The participant may choose whether they join the Calm application vs usual care (questionnaires only) group on a voluntary basis; there is no pre-assignment. The Calm application is a publicly available program that is available to any patient independent of this study.

ELIGIBILITY:
Inclusion Criteria:

Established patients of the Johns Hopkins (JH) Rheumatology Division will be eligible for participation.

* Participants must have one of the following JH rheumatologist-diagnosed and/or confirmed diseases: inflammatory arthritis, scleroderma, myositis, Sjogren's syndrome, systemic lupus erythematosus, and vasculitis.
* Participants must be at least 18 years of age to participate; there is no upper-bound age limit
* Participants must have access to a smartphone or computer to access the Calm app (or webpage) as well as Redcap (which requires an email address) to access the questionnaires

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited | 2 years
  The investigators' goal is to recruit 264 participants. The investigators will report the number of participants recruited which will be a measure of Percentage of target enrollment achieved.
Total number of minutes per participant | 30 days
  The program consists of a total of 150 minutes. The investigators will report the total number of minutes per participant as a measure of adherence to program.

SECONDARY OUTCOMES:
Change in Anxiety as assessed by the Patient Reported Outcomes Measurement Information System (PROMIS) Global-29 profile | Baseline, 30 days
  The PROMIS global-29 measure is reported as a profile. For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured. The anxiety T-score (subscale of PROMIS being used here) ranges from 40-81.
Change in Depression as assessed by the PROMIS Global-29 profile | Baseline, 30 days
  The PROMIS global-29 measure is reported as a profile. For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured. The depression T-score (subscale of PROMIS being used here) ranges from 41-79.
Change in Fatigue as assessed by the PROMIS Global-29 profile | Baseline, 30 days
  The PROMIS global-29 measure is reported as a profile. For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured. The fatigue T-score (subscale of PROMIS being used here) ranges from 33-75.
Change in Physical Function as assessed by the PROMIS Global-29 profile | Baseline, 30 days
  The PROMIS global-29 measure is reported as a profile. For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured. The physical function T-score (subscale of PROMIS being used here) ranges from 22-56.
Change in Social participation as assessed by the PROMIS Global-29 profile | Baseline, 30 days
  The PROMIS global-29 measure is reported as a profile. For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured. The social participation T-score (subscale of PROMIS being used here) ranges from 29-64.
Change in Pain interference as assessed by the PROMIS Global-29 profile | Baseline, 30 days
  The PROMIS global-29 measure is reported as a profile. For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured. The pain interference T-score (subscale of PROMIS being used here) ranges from 41-75.
Change in Sleep disturbance as assessed by the PROMIS Global-29 profile | Baseline, 30 days
  The PROMIS global-29 measure is reported as a profile. For PROMIS instruments, a T-score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured. The sleep disturbance T-score (subscale of PROMIS being used here) ranges from 32-73.
Change in Anxiety as assessed by the PROMIS anxiety computer adaptive testing (CAT) | Baseline, 30 days
  The PROMIS anxiety CAT has a T-score range of 40 to 81. For PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured.
Change in Depression as assessed by the PROMIS depression CAT | Baseline, 30 days
  The PROMIS depression CAT has a T-score range of 38 to 81. For PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured.
Change in Self-Efficacy for managing emotions as assessed by the PROMIS self-efficacy for managing emotions short form (8a) | Baseline, 30 days
  The PROMIS self-efficacy for managing emotions form has a T-score range of 22 to 64. For PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured.
Change in Self-Efficacy for managing symptoms as assessed by the PROMIS self-efficacy for managing symptoms short form (8a) | Baseline, 30 days
  The PROMIS self-efficacy for managing symptoms form has a T-score range of 22 to 63. For PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10. Higher scores indicate more of the trait being measured.
Change in stress as assessed by the Perceived Stress Scale (PSS) | Baseline, 30 days
  The PSS has a score range from 0-40. Higher scores indicate higher perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Dana DiRenzo, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No